CLINICAL TRIAL: NCT01849068
Title: Effects of Selective Inhibition of Cholesterol Absorption With Ezetimibe on Intestinal Cholesterol Homeostasis in Dyslipidemic Men With Insulin-resistance - a Pilot Study
Acronym: EZEmRNA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Patrick Couture, MD, FRCP, PhD, Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INAF-B13-04-1195
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-03

CONDITIONS: Metabolic Syndrome X
MeSH Terms: conditions — Metabolic Syndrome | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ezetimibe (Experimental)
  Interventions: Drug: Ezetimibe
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ezetimibe — Ezetimibe 10 mg/d for 12 weeks
  Other Names: Ezetrol
  Arms: Ezetimibe
Drug: Placebo — Placebo for 12 weeks
  Arms: Placebo

SUMMARY:
Ezetimibe has been shown to inhibit cholesterol absorption and several lines of evidence from in vitro systems and animal models suggest that this effect is associated with an increase in low-density lipoprotein (LDL) receptor expression in the small intestine. The impact of a treatment with ezetimibe on intestinal gene expression and protein mass levels of LDL receptor and other key genes involved in intestinal cholesterol homeostasis will be examined in dyslipidemic men with insulin-resistance. In the present study, gene expression studies and protein mass levels will be assessed on duodenal biopsies by real-time polymerase chain reaction (rt-PCR) and liquid chromatography-mass spectrometry (LC-MS/MS), respectively. The primary objective of this proposal is to examine the effects of ezetimibe on intestinal gene expression (rt-PCR) and protein mass levels (LC-MS/MS) of LDL receptor in dyslipidemic men with insulin-resistance. The secondary objective is to examine the impact of ezetimibe treatment on intestinal gene expression and protein mass levels of sterol regulatory element-binding protein (SREBP)-2, Niemann-Pick C1-Like1 (NPC1L1), ATP binding cassette gene (ABCG)-5/8, proprotein convertase subtilisin/kexin type 9 (PCSK9) and 3-hydroxy-3-methyl-glutaryl-CoA (HMG CoA) reductase.

Primary hypothesis Treatment with ezetimibe 10 mg/day will significantly increase duodenal mRNA and protein mass levels of LDL receptor in dyslipidemic men with insulin-resistance.

Secondary hypothesis Treatment with ezetimibe 10 mg/day will significantly increase duodenal mRNA and protein mass levels of SREBP-2, NPC1L1, ABCG5/8, PCSK9 and HMG CoA reductase in dyslipidemic men with insulin-resistance.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18-60 years
* Waist circumference > 102 cm
* HDL-cholesterol < 1.1 mmol/L
* Triglycerides > 1.7 mmol/L
* Fasting blood glucose > 6.1 mmol/L
* Normal blood pressure (<130/85)

Exclusion Criteria:

* Women
* Men < 18 or > 60 years
* Smokers (> 1 cigarette/day)
* Body weight variation > 10% during the last 6 months prior to the study baseline
* Subjects with a previous history of cardiovascular disease
* Subjects with type 2 diabetes
* Subjects with a monogenic dyslipidemia
* Subjects on hypertension medications or medications known to affect lipoprotein metabolism or the integrity of gastrointestinal mucosa
* Subjects with endocrine or gastrointestinal disorders
* History of alcohol or drug abuse within the past 2 years
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD, FRCP, PhD, Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Ezetimibe First, Then Placebo: First intervention: Ezetimibe 10 mg/d for 12 weeks Second intervention: Placebo for 12 weeks
- Placebo First, Then Ezetimibe: First intervention: Placebo for 12 weeks Second intervention: Ezetimibe 10 mg/d for 12 weeks
Period: Overall Study
Arm/Group | Ezetimibe First, Then Placebo | Placebo First, Then Ezetimibe
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ezetimibe First Then Placebo: First intervention: Ezetimibe 10 mg/d for 12 weeks Second intervention: Placebo 12 weeks
- Placebo First Then Ezetimibe: First intervention: Placebo for 12 weeks Second intervention: Ezetimibe 12 weeks
- Total: Total of all reporting groups
Arm/Group | Ezetimibe First Then Placebo | Placebo First Then Ezetimibe | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.4 (7.9) | 39.4 (13.6) | 39.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Intestinal mRNA Expression Levels of LDL Receptor Between the Two 12-week Interventions
Description: We combined the results at the end of each ezetimibe phase from both sequence (average and standard deviation).
  We combined the results at the end of each placebo phase from both sequence (average and standard deviation).
Time Frame: At the end of the two 12-week interventions (Week 12 and 24)
Measure: Mean (Standard Deviation); unit: #copies/100000 copies housekeeping gene
Groups:
- Ezetimibe: Ezetimibe: Ezetimibe 10 mg/d for 12 weeks Ezetimibe 10 mg/d for 12 weeks
- Placebo: Placebo: Placebo for 12 weeks Placebo for 12 weeks
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 20 | 20
#copies/100000 copies housekeeping gene | 110531 (32604) | 95140 (31840)

2. Secondary Outcome: Change in Intestinal mRNA Expression Levels of SREBP-2, NPC1L1, ABCG5/8, PCSK9 and HMG CoA Reductase Between the Two 12-week Interventions
Description: as for outcome 1
Time Frame: At the end of the two 12-week interventions (Week 12 and 24)
Measure: Mean (Standard Deviation); unit: #copies/100000 copies housekeeping gene
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 20 | 20
#copies/100000 copies housekeeping gene
  HMGCoA reductase | 354911 (102607) | 311268 (88237)
  PCSK9 | 9079 (5816) | 8091 (6131)
  SREBP-2 | 193012 (32787) | 182349 (36681)
  NPC1L1 | 454298 (97707) | 448686 (138746)
  ABCG5 | 271811 (111688) | 283863 (132434)
  ABCG8 | 125315 (46842) | 129551 (63246)

3. Secondary Outcome: Change in Intestinal Protein Levels of LDL Receptor Between the Two 12-week Interventions
Description: as for outcome 1
Time Frame: At the end of the two 12-week interventions (Week 12 and 24)
Population: Data will never be analyzed because the mRNA expression of LDL receptor is sufficient.
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Protein Levels of SREBP-2, NPC1L1, ABCG5/8, PCSK9 and HMG CoA Reductase Between the Two 12-week Interventions
Description: as for outcome 1
Time Frame: At the end of the two 12-week interventions (Week 12 and 24)
Population: Data will never be analyzed because the mRNA expression of SREBP-2, NPC1L1, ABCG5/8, PCSK9 and HMG CoA reductase are sufficient.
Arm/Group | Ezetimibe | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Ezetimibe: Ezetimibe 10 mg/d for 12 weeks Ezetimibe 10 mg/d for 12 weeks
- Placebo: Placebo for 12 weeks Placebo for 12 weeks
Arm/Group | Ezetimibe | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No